CLINICAL TRIAL: NCT04622462
Title: A Multi-Centre Prospective Community-Based Observational Study on Prediction of Malignant Progression of Clinically Suspicious Oral Lesions with STRATICYTE
Brief Title: Early Prediction of Oral Cancer by S100A7 Immunohistochemistry Signature-based Assessment
Status: Recruiting | Type: Observational
Sponsor: Proteocyte Diagnostics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-STR-PPOEL-1
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Oral Neoplasm
Keywords: Leukoplakia; Erythroplakia; Erythroleukoplakia; Lesion; Oral Epithelial Dysplasia; S100A7 Biomarker; S100A7 Immunohistochemistry Signature-based; Early Diagnosis; STRATICYTE; Oral Neoplasia; Oral Epithelial Atypia; Hyperplasia; Hyperkeratosis; Oral Squamous Cell Carcinoma; Oral Cancer; Potentially Premalignant Oral Epithelial Lesion; OPMD; Mild Dysplasia; Moderate Dysplasia; Severe Dysplasia; Low-grade Dysplasia; High-grade Dysplasia; Personalized Medicine; Predictive Assay; Whole Slide Imaging; Computational Pathology; Digital Pathology; Artificial Intelligence; Machine Learning; OPML; Oral Potentially Malignant Disorder; Oral Potentially Malignant Lesion
MeSH Terms: conditions — Mouth Neoplasms; Leukoplakia; Erythroplasia; Disease; Hyperplasia; Keratoderma, Palmoplantar, Epidermolytic; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Formalin-fixed paraffin-embedded tissue sections stained with H&E and S100A7
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Oral Mucosal Biopsies With or Without Evidence of Epithelial Dysplasia: No evidence of dysplasia
  Mild dysplasia
  Moderate dysplasia
  Severe dysplasia
  Interventions: Procedure: Standard of Care Histopathology; Procedure: STRATICYTE Assessment

INTERVENTIONS:
Procedure: Standard of Care Histopathology — Assessment for mild, moderate, or severe dysplasia, and risk of progression to oral cancer
  Other Names: H&E assessment for dysplasia grade
Procedure: STRATICYTE Assessment — Assessment for risk of progression to oral cancer
  Other Names: S100A7 Immunohistochemistry Signature-based Assessment

SUMMARY:
The purpose of this observational study is to evaluate the utility of the S100A7 immunohistochemistry signature-based assessment - STRATICYTE - in determining the risk of progression to cancer of clinically suspicious oral lesions.

DETAILED DESCRIPTION:
Background: The standard of care for potentially premalignant oral epithelial lesion (PPOEL) risk assessment for progression to cancer is dysplasia grading by histopathology. With significant overlap between dysplasia grades and high inter- and intra-observer variations, dysplasia grading alone has been shown to be inadequate as a prognostic tool. To investigate the utility of the S100A7 immunohistochemistry signature-based assessment - STRATICYTE - in the early diagnosis of invasive oral cancer, a prospective multi-center observational study was designed with specimens obtained from community-based practices.

Methods: Patients that qualify to enroll in the study will be assessed for both standard of care histopathological assessment for dysplasia grade and STRATICYTE risk assessment, and followed for up to 60 months (from initial biopsy) to determine the outcome of their oral lesion(s).

ELIGIBILITY:
Inclusion Criteria:

* Any clinically suspicious lesion biopsied to rule-out oral epithelial dysplasia/oral squamous cell carcinoma

Exclusion Criteria:

* Biopsied lesion with or without dysplasia concomitant with oral squamous cell carcinoma at initial biopsy

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be selected from community-based Oral & Maxillofacial Surgery practices in the provinces of Ontario and Alberta, Canada
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-03-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Malignant Transformation Rate: Dysplasia | 60 months
  Cancer progression rate in patients with oral neoplasia with dysplasia and STRATICYTE Low-Risk or Elevated Risk

SECONDARY OUTCOMES:
Malignant Transformation Rate: No Dysplasia | 60 months
  Cancer progression rate in patients with oral neoplasia without dysplasia and STRATICYTE Low-Risk or Elevated-Risk
Recurrence Rate | 60 months
  Recurrence rate in patients with oral neoplasia with or without dysplasia and STRATICYTE Low-Risk or Elevated-Risk

CONTACTS AND LOCATIONS:
Overall Officials: Mark Darling, MSc, MChD, Principal Investigator — Western University
Locations (3):
- Canada (3):
  - Kingsway Oral & Maxillofacial Surgery, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Western University, London, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hwang JTK, Dammling C, McCord C, McGuire T, Park EP, Filkowski J, Shaw E, McMullen S, Nwigwe A, Ekwaru JP, McGaw WT, Lung KE, Seikaly H, Renick B, Lin DM, Morlandt A, Pritzker KH, Darling MR. External Validation of Straticyte, a Quantitative Biomarker-Based Risk Assay in Predicting Oral Cancer. J Maxillofac Oral Surg. 2025 Oct;24(5):1351-1357. doi: 10.1007/s12663-024-02362-7. Epub 2024 Oct 29. PMID 41054469
- [Background] Hwang JT, Gu YR, Shen M, Ralhan R, Walfish PG, Pritzker KP, Mock D. Individualized five-year risk assessment for oral premalignant lesion progression to cancer. Oral Surg Oral Med Oral Pathol Oral Radiol. 2017 Mar;123(3):374-381. doi: 10.1016/j.oooo.2016.11.004. Epub 2016 Nov 22. PMID 28110942
- [Background] Kaur J, Matta A, Kak I, Srivastava G, Assi J, Leong I, Witterick I, Colgan TJ, Macmillan C, Siu KW, Walfish PG, Ralhan R. S100A7 overexpression is a predictive marker for high risk of malignant transformation in oral dysplasia. Int J Cancer. 2014 Mar 15;134(6):1379-88. doi: 10.1002/ijc.28473. Epub 2013 Oct 8. PMID 24122701
- [Background] Tripathi SC, Matta A, Kaur J, Grigull J, Chauhan SS, Thakar A, Shukla NK, Duggal R, DattaGupta S, Ralhan R, Siu KW. Nuclear S100A7 is associated with poor prognosis in head and neck cancer. PLoS One. 2010 Aug 3;5(8):e11939. doi: 10.1371/journal.pone.0011939. PMID 20689826
- [Background] Ralhan R, Desouza LV, Matta A, Tripathi SC, Ghanny S, Dattagupta S, Thakar A, Chauhan SS, Siu KW. iTRAQ-multidimensional liquid chromatography and tandem mass spectrometry-based identification of potential biomarkers of oral epithelial dysplasia and novel networks between inflammation and premalignancy. J Proteome Res. 2009 Jan;8(1):300-9. doi: 10.1021/pr800501j. PMID 19072117
- [Background] Ralhan R, Desouza LV, Matta A, Tripathi SC, Ghanny S, Datta Gupta S, Bahadur S, Siu KW. Discovery and verification of head-and-neck cancer biomarkers by differential protein expression analysis using iTRAQ labeling, multidimensional liquid chromatography, and tandem mass spectrometry. Mol Cell Proteomics. 2008 Jun;7(6):1162-73. doi: 10.1074/mcp.M700500-MCP200. Epub 2008 Mar 13. PMID 18339795